CLINICAL TRIAL: NCT05980325
Title: Exercise for Fighting Oncology Repercussions After Treatment: the EFFORT Trial
Brief Title: Exercise for Fighting Oncology Repercussions After Treatment
Acronym: EFFORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Col·legi de Fisioterapeutes de Catalunya (Unknown); Ajuntament de Mataró (Unknown)
Responsible Party: Principal Investigator, Raquel Sebio, Senior Lecturer, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCM-EFFORTv3
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
Keywords: Neoplasms; Exercise Therapy; Side Effects; Cancer-related Fatigue; Quality of Life
MeSH Terms: conditions — Neoplasms | interventions — Nordic Walking; Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nordic Walking (Experimental): Patients in this arm will be assigned to a 12-week exercise intervention twice weekly based on Nordic Walking (NW). The intervention will be structured as follows: i) 10 min warm-up, ii) 40 min NW with muscle strengthening exercises interspersed in between and iii) 10 min cool-down. Intensity will be monitored with a heart rate monitor (when available) and/or Borg Scale to reach a moderate intensity for the first 6 weeks (4 - 6 or 55-65% HR reserve) to a moderate-to-high intensity the following weeks (7 - 8 or 65-75% HR reserve).
  Interventions: Behavioral: Nordic Walking
- Aquatic Exercise (Experimental): Patients in this group will be assigned to a 12-week, twice weekly water-based exercise programme to be conducted at a chest-high swimming pool kept around 30 to 32 degrees Celsius. Each session will be structured as previous: i) 10 min warm up; ii) 40 min of combined endurance and strength exercise training and iii) 10 min cool down. Intensity will be monitored using the Borg Scale to be moderate during the first 6 weeks (4 - 6) and moderate-to-high the following 6 weeks (7-8).
  Interventions: Behavioral: Aquatic Exercise
- Functional Exercise Training (Active Comparator): In this group, patients will participate in a traditional, circuit-based exercise training at a fitness facility twice daily during 12 weeks. Each session will consist of: i) 10 min warm up; ii) 40 min of combined resistance and endurance training using a circuit-based structure and iii) 10 min cool-down. Intensity will be monitored with a HR monitor (when available) and/or Borg Scale to reach a moderate intensity for the first 6 weeks (4 - 6 or 55-65% HR reserve) and will progress to moderate-to-high over the following weeks (7-8 or 65-75% HR reserve).
  Interventions: Behavioral: Functional Exercise Training

INTERVENTIONS:
Behavioral: Nordic Walking — A 12-week Nordic Walking exercise programme supervised twice weekly
  Arms: Nordic Walking
Behavioral: Aquatic Exercise — A 12-week water-based exercise training programme supervised twice weekly
  Arms: Aquatic Exercise
Behavioral: Functional Exercise Training — A 12-week circuit-based exercise training programme supervised twice weekly
  Arms: Functional Exercise Training

SUMMARY:
Cancer survival rates are currently on the verge of 70% at 5 years since diagnosis. Recent improvements in main cancer therapies including chemotherapy, radiotherapy, surgery and immunotherapy as well as developments of new biological therapies have significantly improved survival rates but unfortunately, cancer-related side effects continue to affect many patients even years after completion of main treatments. Exercise has been shown to not only ameliorate cancer-related effects before, during and after treatment but also improve disease-free and overall survival rates by decreasing risk factors associated with cancer risk and improving resilience to treatment. In this non-randomised, three-arm study, we aim to assess the effects of three forms of exercise (i.e: Nordic Walking, Aquatic Exercise and Functional Exercise) on physical performance, cancer-related fatigue, health-related quality of life and cancer-specific symptoms in a wide range of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with cancer
* Completion of any cancer therapy in the previous 3 months with the exception of hormonal therapy
* Patients living within the Maresme Area
* No contraindications for exercise (oncology clearance or Physical Activity Readiness Questionnaire negative)

Exclusion Criteria:

* Patients with any neurologic, cognitive or musculoskeletal impairments that prevent them to engage in any assessment test or exercise modality.
* Patients with unstable cardiac, respiratory or metabolic diseases
* Unable to speak or read Catalan or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | 12 weeks from baseline
  HRQoL measured with the EORTC Quality of Life C30 questionnaire

SECONDARY OUTCOMES:
Cancer-related fatigue | 12 weeks from baseline
  Cancer-related fatigue as measure with the Brief Fatigue Inventory
Cardiorespiratory fitness | 12 weeks from baseline
  A steady state cardiopulmonary exercise testing with breath-by-breath analysis and lactate measurement to determine submaximal cardiorespiratory fitness
Estimated one-repetition maximum | 12 weeks from baseline
  Estimated maximal muscle strength using a linear Encoder for two main muscle groups: i) chest and ii) quads
Lower limb muscle endurance | 12 weeks from baseline
  Lower limb muscle endurance measured as the maximum number of sit-to-stand repetitions performed in 30 seconds
Functional capacity | 12 weeks from baseline
  Walking distance covered during a self-pace 6 minute walk test

IPD SHARING:
Plan to Share IPD: No